CLINICAL TRIAL: NCT04546984
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Ascending Multiple Doses to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics，and Randomized, Open-label，Crossover, Food Effect Study of HEC96719 in Healthy Chinese Subjects
Brief Title: Multiple Dose Safety, Tolerability, PK，PD and Food Effect Study of HEC96719 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC96719-P-02/CRC-C2028
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single dose of HEC96719 （Part 1，Fed/Fasting） (Experimental): Following an overnight fast of at least 10 hours, a single dose of HEC96719 will be administered on 2 separate occasions (fasting and after meal) in a randomized crossover fashion with different food restrictions.
  Interventions: Drug: HEC96719
- Mulltiple doses HEC96719（ Part 2, Cohort 1） (Experimental): Healthy subjects receive multiple doses of HEC96719 or matching placebo
  Interventions: Drug: HEC96719
- Mulltiple doses HEC96719（ Part 2, Cohort 2） (Experimental): Healthy subjects receive multiple doses of HEC96719 or matching placebo
  Interventions: Drug: HEC96719
- Mulltiple doses HEC96719（ Part 2, Cohort 3） (Experimental): Healthy subjects receive multiple doses of HEC96719 or matching placebo
  Interventions: Drug: HEC96719
- Mulltiple doses HEC96719（ Part 2, Cohort 4） (Experimental): Healthy subjects receive multiple doses of HEC96719 or matching placebo
  Interventions: Drug: HEC96719
- Mulltiple doses HEC96719（ Part 2, Cohort 5） (Experimental): Healthy subjects receive multiple doses of HEC96719 or matching placebo
  Interventions: Drug: HEC96719

INTERVENTIONS:
Drug: HEC96719 — Part 2：Mulltiple doses up to 10 days

SUMMARY:
The Safety, Tolerability, Pharmacokinetic, Pharmacodynamics and Food Effect Study of HEC96719 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study, able to understand and sign the informed consent, and able to complete the the study in accordance with the requirements of the study.
* Female subjects who are not pregnant or lactating and male subjects whose female partners are fertile shall voluntarily take effective contraceptive measures from the date of signing the informed consent form to 3 months after the medication.
* When signing the informed consent, 18 years old ≤the age≤45 years old(including the critical value), gender is not limited.
* Male body weight ≥50kg, female body weight ≥45kg, and body mass index (BMI) in the range of 18-28 kg/m2 (including the critical value).
* No clinical significance of vital signs, physical examination, laboratory examination, electrocardiogram, ultrasound abdomen and chest X-ray (posterior and anterior) results.

Exclusion Criteria:

* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis.
* Those who are known to have allergy history or allergy constitution to the test preparation and any of its components or related preparations.
* Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
* Positive results from urine drug screen test.
* Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
* Subjects who plan to receive or have had organ transplants.
* Subjects considered by the investigator to have other factors unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of HEC96719 by Assessment of the Number of Adverse Events | up to 17 days
  To investigate the safety and tolerability of HEC96719 by assessment of AEs (non-serious and serious) following administration of oral solution in MAD

SECONDARY OUTCOMES:
Cmax | up to 96 hours
  Maximum Plasma Concentration(Cmax)of HEC96719
AUC | up to 96 hours
  Area Under the Curve(AUC) of HEC96719
Tmax | up to 96 hours
  Maximum Peak Time(Tmax) of HEC96719
T1/2 | up to 96 hours
  Maximum Peak Time(Tmax) of HEC96719

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai xuhui district central hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No